CLINICAL TRIAL: NCT03196973
Title: A Phase III, Multicenter, Randomized, Double-Blind Clinical Trial to Assess the Efficacy and Safety of DF289 Plus DF277 Otic Solution Compared to DF289 Otic Solution and to DF277 Otic Solution in the Treatment of Acute Otitis Externa (AOE)
Brief Title: Efficacy and Safety of DF289 Plus DF277 Otic Solution in the Treatment of Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DF289OT3-16IA01
Record Dates: First submitted 2017-06-16; First posted 2017-06-23 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-11

CONDITIONS: Acute Otitis Externa
MeSH Terms: interventions — Anti-Bacterial Agents; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DF289 plus DF277 (Experimental): Otic solution
  Interventions: Drug: DF289 plus DF277
- DF289 (Active Comparator): Otic solution
  Interventions: Drug: DF289
- DF277 (Active Comparator): Otic solution
  Interventions: Drug: DF277

INTERVENTIONS:
Drug: DF289 plus DF277 — 1 vial into the affected ear twice daily for 7 days
  Other Names: Antibiotic and Corticosteroid
  Arms: DF289 plus DF277
Drug: DF289 — 1 vial into the affected ear twice daily for 7 days
  Other Names: Antibiotic
  Arms: DF289
Drug: DF277 — 1 vial into the affected ear twice daily for 7 days
  Other Names: Corticosteroid
  Arms: DF277

SUMMARY:
The purpose of this study is to determine if a combination of an antibiotic plus a corticosteroid is safe and effective in treating AOE

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated AOE of less tan 21 days, defined as a total symptom score of at least 2 for otalgia, 2 for edema and 1 for otorrhea
* Brighton Grading of II or III
* Culture-based diagnosis of acute bacterial otitis externa
* Willingness to refrain from swimming through end of the study

Exclusion Criteria:

* Previous episode of AOE within 4 weeks prior to enrollment, or 2 or more episodes of AOE within 6 months prior to the enrollment.
* Tympanic membrane perforation
* Any condition or situation likely to cause the patient to be unable or unwilling to comply with study treatment or attend all study visits
* Any condition in the patient or parent/guardian that, in the judgment of the principal investigator, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Jiménez, Study Director — Salvat
Locations (1):
- Laboratorios SALVAT, Esplugues de Llobregat, Spain

REFERENCES:
- [Derived] Chu L, Acosta AM, Aazami H, Dennis P, De Valle O, Ehmer D Jr, Hedrick JA, Ansley JF. Efficacy and Safety of Ciprofloxacin Plus Fluocinolone Acetonide Among Patients With Acute Otitis Externa: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2221699. doi: 10.1001/jamanetworkopen.2022.21699. PMID 35834251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DF289 Plus DF277 | DF289 | DF277
Started | 197 | 196 | 100
Completed | 188 | 184 | 95
Not Completed | 9 | 12 | 5
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Lack of Efficacy | 2 | 6 | 1
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — Consent withdrawn | 2 | 1 | 0
Not completed — Administration of a wrong kit of study medication | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: CITT Population (Randomized patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | DF289 Plus DF277 | DF289 | DF277 | Total
Number analyzed (Participants) | 197 | 196 | 100 | 493
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 57 | 31 | 145
  Between 18 and 65 years | 102 | 115 | 54 | 271
  >=65 years | 38 | 24 | 15 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (23.81) | 38.4 (22.64) | 38.7 (22.79) | 38.2 (23.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 101 | 56 | 254
  Male | 100 | 95 | 44 | 239
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 29 | 30 | 15 | 74
  White | 162 | 161 | 82 | 405
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 2 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 197 | 196 | 100 | 493

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Cure (Clinical + Microbiological Cure)
Description: Therapeutic cure will be considered achieved if edema, otalgia and otorrhea are resolved with no further requirement of antimicrobial therapy and bacteriological response is Eradication or Presumed Eradication
Time Frame: End of Treatment (Day 8+2)
Population: Randomized patients with positive culture for pathogens at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | DF289 Plus DF277 | DF289 | DF277
Number analyzed (Participants) | 103 | 91 | 45
Participants | 63 | 49 | 20

2. Secondary Outcome: Time to End of Pain
Description: First day on which there is no use of analgesics, the pain score is zero and remains zero until end of study
Time Frame: From baseline to End of Study (Day 15+2)
Population: Randomized patients with positive culture for pathogens at baseline
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DF289 Plus DF277 | DF289 | DF277
Number analyzed (Participants) | 103 | 91 | 45
days | 5.0 [4.23 to 6.34] | 5.9 [4.26 to 7.25] | 7.7 [6.74 to 9.00]

ADVERSE EVENTS:
Time Frame: From study entry to Visit 4(Day 15+2)
Description: Related and unrelated adverse events are reported which frequency was 1% or more in one of the arms.
  2 subjects (1 from the DF289Plus DF277 arm and 1 from the DF289) are excluded from the safety population because they did not receive any dose of study medication.
Arm/Group | DF289 Plus DF277 | DF289 | DF277
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/195 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/196 | 0/195 | 0/100
Other Adverse Events (participants affected / at risk) | 11/196 | 12/195 | 4/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DF289 Plus DF277 (N=196) | DF289 (N=195) | DF277 (N=100)
Acute Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — The SAE was not related to the study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DF289 Plus DF277 (N=196) | DF289 (N=195) | DF277 (N=100)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 0 (0)
ear pruritus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
application site pain (General disorders) | 4 (4) | 0 (0) | 0 (0)
cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 4 (4) | 6 (6) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication by PI of the Study Results shall not be made before the first multi-center publication.

PI shall allow Sponsor not less than 60 days to review any manuscript and not less than 30 days to review any other documentation which describes or discloses the Study Results. Sponsor can request an additional 60 days.

Sponsor reserves the right to remove all Confidential Information from any publications or presentations.

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT03196973/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT03196973/SAP_002.pdf